CLINICAL TRIAL: NCT03752502
Title: Effects of Cerebral and Peripheral Electrical Stimulation on Conditioned Pain Modulation in Healthy Subjects.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidade Federal do Piauí (Other)
Responsible Party: Principal Investigator, Fuad Ahmad Hazime, Assistant Professor - Physical Therapy Department, Universidade Federal do Piauí
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1.584.966
Record Dates: First submitted 2018-11-21; First posted 2018-11-26 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cerebral stimulation (Experimental): Active transcranial direct current stimulation
  tDCS: 20 minutes, 2mA, primary motor cortex anode (contralateral to the lesion) and supraorbital cathode (ipsilateral to the lesion).
  Interventions: Procedure: Transcranial direct current stimulation (tDCS)
- Combined stimulation (Experimental): Active transcranial direct current stimulation combined with active peripheral electrical stimulation (PES)
  tDCS: 20 minutes, 2mA, primary motor cortex anode (contralateral to the lesion) and supraorbital cathode (ipsilateral to the lesion).
  PES: 20 minutes, 10Hz (frequency), 100µs (pulse duration), intensity at sensorial level.
  Interventions: Procedure: Transcranial direct current stimulation (tDCS); Procedure: Peripheral electrical stimulation (PES)
- Sham cerebral stimulation (Sham Comparator): Sham transcranial direct current stimulation combined with active peripheral electrical stimulation (PES)
  tDCS: 20 minutes (30s ON), 2mA, primary motor cortex anode (contralateral to the lesion) and supraorbital cathode (ipsilateral to the lesion).
  Interventions: Procedure: Sham tDCS
- Peripheral stimulation (Experimental): Active peripheral electrical stimulation (PES).
  PES: 20 minutes, 10Hz (frequency), 100µs (pulse duration), intensity at sensorial level.
  Interventions: Procedure: Peripheral electrical stimulation (PES); Procedure: Sham tDCS

INTERVENTIONS:
Procedure: Transcranial direct current stimulation (tDCS) — Transcranial direct current stimulation (tDCS) is a noninvasive brain stimulation (NIBS) technique that has been investigated for the management of various chronic pain conditions. However, as a monotherapy for pain relief, this therapy still has controversial results.
  Arms: Cerebral stimulation; Combined stimulation
Procedure: Peripheral electrical stimulation (PES) — Peripheral electrical stimulation (PES) activates a complex neural network involving a series of neurotransmitters and receptors capable of promoting segmental and extrasegmental analgesia.
  Arms: Combined stimulation; Peripheral stimulation
Procedure: Sham tDCS — Transcranial direct current stimulation (tDCS) is a noninvasive brain stimulation (NIBS) technique that has been investigated for the management of various chronic pain conditions. However, as a monotherapy for pain relief, this therapy still has controversial results.
  Arms: Peripheral stimulation; Sham cerebral stimulation

SUMMARY:
The Neuromatrix pain model and new findings on pain chronification process point to a greater efficacy of treatments that address central and peripheral rather than only peripheral structures. Both cerebral and peripheral electrical stimulations can modulate brain areas involved in pain processing. However, their effects on pain modulation systems and clinical outcomes are lacking.

This study aims to investigate the efficacy of transcranial direct current stimulation (tDCS) and peripheral electrical stimulation (PES) alone as well tDCS combined with PES on pressure pain threshold and conditioned pain modulation in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects without medical complaints.

Exclusion Criteria:

Concurrent medication likely to affect cognitive performance pregnancy or possible pregnancy history of drug or alcohol abuse or dependence recent head injury (in the last 3 months) history of seizure or stroke.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2021-11-27 (Actual)

PRIMARY OUTCOMES:
Pressure pain threshold | Pre and Post-test (immediately after tDCS)
  Pressure pain threshold (PPT) is defined as the minimum force applied which induces pain.
Conditioned pain modulation | Pre and Post-test (immediately after tDCS)
  Conditioned pain modulation paradigms consist of the evaluation of a painful test stimulus followed by a second evaluation either at the same time as a distant, painful conditioning stimulus.
  PPT will be evaluated following a conditioning stimulus condition (hand immersion in a cold water).

OTHER OUTCOMES:
Anxiety | Pre-test (before tDCS)
  Visual analogue scale (VAS) for anxiety assesses anxiety symptoms that we tracked as possible confounding factor.
  The VAS for general anxiety is assessed by a horizontal 100-mm-long line. The extreme left end points to no anxiety, and the extreme right end to the worst anxiety possible.
Depression | Pre-test (before tDCS)
  Beck depression inventory (BDI) for depressive symptoms that we tracked as possible confounding factor.
  The BDI is a tool of self-assessment of depression using a questionnaire with 21 items whose intensity varies from 0 to 3 (higher scores indicating more depressive symptoms).
Pain catastrophizing | Pre-test (before tDCS)
  Catastrophizing pain scale that we tracked as possible confounding factor.
  The pain catastrophizing scale consists of 13 sentences describing pain-related thoughts or feelings. These are divided into 3 domains: rumination, magnification and helplessness.
  The total score on the questionnaire can lie between 0 - 52 where a higher score indicates higher levels of pain catastrophizing thoughts.

CONTACTS AND LOCATIONS:
Overall Officials: Fuad Hazime, PhD, Principal Investigator — Federal University of Piaui
Locations (1):
- Department of Physical Therapy. Federal University of Piaui, Parnaíba, Piauí, Brazil